CLINICAL TRIAL: NCT01857674
Title: Evaluation of Laryngeal Ultrasonography Performance in Predicting Major Post Extubation Laryngeal Edema in Intensive Care Patients
Acronym: ECHOLPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00141-44
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-05

CONDITIONS: Laryngeal Edema; Acute Respiratory Failure Requiring Reintubation
Keywords: Laryngeal edema; Post-extubation; Acute respiratory distress; Ultrasonography; Intensive care unit
MeSH Terms: conditions — Laryngeal Edema; Acute Lung Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* For patient in intensive care unit, extubation failure is defined as the necessity of early reintubation after scheduled extubation, with Increased morbidity and mortality, so it seems important to quickly identify patients with high risk of post-extubation acute respiratory failure.
* Major post-extubation laryngeal edema is one of extubation failure causes, and its incidence vary in literature from 4 to 37%.
* We can't currently predict arising of a major post-extubation laryngeal edema. However, a recent pilot study showed that laryngeal ultrasonography could help to identify patients with high risk of post-extubation stridor, measuring ultrasonic leak volume and cuff-deflated air-column width, of which we propose to assess diagnostic performance.

DETAILED DESCRIPTION:
Definitions:

Intubation is a traumatism for laryngeal mucous membrane. Due to local inflammatory reaction, laryngeal edema occurs in nearly all intubated patients, but only some of them develop clinical symptoms, as post-extubation stridor or acute respiratory distress. Stridor is commonly defined as a high-pitched sound produced by airflow through a narrowed airway, and accepted as a clinical marker of post-extubation laryngeal edema. The main complication of post-extubation laryngeal edema is reintubation, defining major post-extubation laryngeal edema. Early recognition of laryngeal edema is essential since these patients have the highest risk of evolving to respiratory distress and extubation failure. Even before extubation, signs indicative of laryngeal edema may be present. The search for a test that adequately identifies patients at risk for extubation failure is ongoing.

Trial Procedures:

* At day 0: Selection of patients filling inclusion criteria. Oral and written information of patient and his refer person, and collecting of non-opposition.
* At day 0: inclusion of patients ventilated with inspiratory assistance just before schedulded extubation. Information of patient on procedure course.
* First ultrasonography of protocol: The patient is in the supine position, with the neck hyper-extended, and the probe is placed on cricothyroid membrane with a transverse view of the larynx. The standard scanning plane is predetermined: it should contain several landmarks, including the vocal cords, false cords, thyroid cartilage and arytenoids cartilage. The oral and laryngeal secretions are suctioned. Ultrasonic air-leak volume is defined by difference between air-column width cuff inflated and air-column width cuff deflated. Shape of air-column cuff inflated and cuff deflated is also recorded in observation notebook.
* Then the patient is extubated after spontaneous ventilation trial, according to unit protocol, by the physician in charge. After extubation, surveillance of post-extubation stridor and acute respiratory distress occurrence during the first 24 hours.
* If the patient is reintubated for major post-extubation laryngeal edema, onset of 48 hours corticotherapy, and realization of second, third and fourth laryngeal ultrasonography, daily to next schedulded extubation.
* At discharge of intensive care unit, data collection about mechanical ventilation duration, intensive care hospitalization duration, occurrence of ventilation-acquired pneumopathy, mortality at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Intubated and ventilated for more than 48 hours.
* Filling mechanical ventilation weaning criteria according to the 6th consensus conference on intensive care medicine.
* Affiliated to French Sociale Sécurity.

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Under 18 or under guardianship patients
* Laryngeal pathology: benign or malignant tumor, unilateral or bilateral paralysis of recurrent laryngeal nerve, laryngitis
* Past history of cervical surgery or radiotherapy
* Technical impossibility of laryngeal ultrasonography: wound or locale infection in ultrasonic plan
* Self-extubation or accidental extubation
* Refusal to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Adults were admitted to the surgical (20 beds) and medical (20 beds)intensive care unit of besançon University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Performance of laryngeal ultrasonography in predicting major post extubation laryngeal edema in intensive care patients. | Within the first 24 hours after extubation
  Sensitivity, specificity, positive predictive value and negative predictive value of ultrasonic air-leak volume in predicting major post-extubation laryngeal edema in intensive care patients.
  A post-extubation laryngeal edema is major when inducing acute respiratory failure requiring early reintubation.
  We assume that, among patients with post-extubation laryngeal edema,the ultrasonic air-leak volume is lower than among patients without post-extubation laryngeal edema.

SECONDARY OUTCOMES:
Performance of laryngeal ultrasonography in predicting post-extubation stridor in intensive care patients. | Within the first 24 hours after extubation
  Sensitivity, specificity, positive predictive value and negative predictive value of ultrasonic air-leak volume in predicting post-extubation stridor.
  Post-extubation stridor is commonly defined as a high-pitched sound produced by airflow through a narrowed airway, and is accepted as a clinical marker of laryngeal edema following extubation. So stridor is widely used as outcome measure for post-extubation laryngeal edema.
Frequency of major post-extubation laryngeal edema and post-extubation stridor | Within the first 24 hours after extubation
  In literature, incidence of post-extubation stridor is from 2 to 15%, and incidence of major post-extubation laryngeal edema is from 4 to 37%. We would confront incidence of post-extubation laryngeal edema in our cohort and in literature.
Risk factors of major post-extubation laryngeal edema in intensive care unit | From ICU admission to day of inclusion
  Several studies have identified risk factor for post-extubation laryngeal edema, but controversy remains.
Evolution of ultrasonic parameters with corticotherapy after reintubation for a major post-extubation laryngeal edema | Daily from day 1 to day 3 after reintubation for a major post-extubation laryngeal edema
  The recommended treatment of major post-extubation laryngeal edema is corticotherapy during 48 hours. By an anti-inflammatory effect, the swelling of laryngeal area decreases under corticoids, so we assume that there is a modification of ultrasonic parameters values during this period.
Evaluation of impact of major post-extubation laryngeal edema occurence on mechanical ventilation duration, hospitalization duration and mortality in intensive care unit | Within 28 days after inclusion in study
  Occurence of major post-extubation laryngeal edema leads to increase morbidity and mortality because of reintubation and its complications. In our cohort, some patients would need to be reintubate, others don't, so we would confront data between these 2 groups.
Inter-observer reproductibility of ultrasound scanning and ultrasonic air-leak volume measurement | Day 1 of inclusion
  In first 100 included patients,we would perform 2 laryngeal ultrasonograpy to assess inter-observer reproductibility of this new test.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Besançon, Besançon, France

REFERENCES:
- [Background] Ding LW, Wang HC, Wu HD, Chang CJ, Yang PC. Laryngeal ultrasound: a useful method in predicting post-extubation stridor. A pilot study. Eur Respir J. 2006 Feb;27(2):384-9. doi: 10.1183/09031936.06.00029605. PMID 16452597
- [Background] Wittekamp BH, van Mook WN, Tjan DH, Zwaveling JH, Bergmans DC. Clinical review: post-extubation laryngeal edema and extubation failure in critically ill adult patients. Crit Care. 2009;13(6):233. doi: 10.1186/cc8142. Epub 2009 Dec 1. PMID 20017891
- [Background] Sustic A. Role of ultrasound in the airway management of critically ill patients. Crit Care Med. 2007 May;35(5 Suppl):S173-7. doi: 10.1097/01.CCM.0000260628.88402.8A. PMID 17446776
- [Background] Frutos-Vivar F, Esteban A, Apezteguia C, Gonzalez M, Arabi Y, Restrepo MI, Gordo F, Santos C, Alhashemi JA, Perez F, Penuelas O, Anzueto A. Outcome of reintubated patients after scheduled extubation. J Crit Care. 2011 Oct;26(5):502-509. doi: 10.1016/j.jcrc.2010.12.015. Epub 2011 Mar 3. PMID 21376523